CLINICAL TRIAL: NCT06105203
Title: A Multicenter Randomized Clinical Trial to Assess the Advantages of Robotic Total Mesorectal Excision in Preserving External Sphincter in Patients with Middle and Low Rectal Cancer.
Brief Title: RATME Vs LATME in Middle and Low Rectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Jilin Provincial Tumor Hospital (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STARS-RC05
Record Dates: First submitted 2023-09-03; First posted 2023-10-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Total Mesorectal Excision; Rectal Neoplasms; Robotic Surgical Procedures; Laparoscopy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RATME (Other): In RaTME groups, the low anterior resection and TME was finished with the assistance of robot (da Vinci Xi surgical system)
  Interventions: Procedure: Robotic-assisted total mesorectal excision
- LATME (Other): In LaTME groups, the low anterior resection and mesorectal excision procedures was completed under laparoscopy.
  Interventions: Procedure: laparoscopic-assisted total mesorectal excision

INTERVENTIONS:
Procedure: Robotic-assisted total mesorectal excision — TME will be performed with the assistance of robot in rectal cancer
  Arms: RATME
Procedure: laparoscopic-assisted total mesorectal excision — TME will be performed with the assistance of laparoscopy in rectal cancer
  Arms: LATME

SUMMARY:
This is a multicenter, superior, randomized controlled trial designed to compare Robotic-assisted total mesorectal excision (RATME) and laparoscopic-assisted total mesorectal excision (LATME) for middle and low rectal cancer. The primary endpoint is the incidence of intersphincteric resection (ISR). The secondary outcomes are coloanal anastomosis (CAA), conversion to open, conversion to transanal TME (TaTME), incidence of abdominoperineal resection (APR), postoperative morbidity and mortality within 30 days after surgery, pathological outcomes, long-term survival outcomes, functional outcomes, and quality of life.

DETAILED DESCRIPTION:
Robotic-assisted total mesorectal excision (RATME) has been gradually applied by colorectal surgeons. Most surgeons consider RATME a safe method and believe it can facilitate total mesorectal excision (TME) in rectal cancer, especially middle and low rectal cancer with a narrow pelvis. Therefore, this trial investigates whether RATME has technical advantages and increase intersphincteric resection rate compared with laparoscopic-assisted TME (LATME) in middle and low rectal cancer.

This is a multicenter, superior, randomized controlled trial designed to compare RATME and LATME for middle and low rectal cancer. The primary endpoint is the incidence of intersphincteric resection (ISR). The secondary outcomes are coloanal anastomosis (CAA), conversion to open, conversion to transanal TME (TaTME), incidence of abdominoperineal resection (APR), postoperative morbidity and mortality within 30 days after surgery, pathological outcomes, long-term survival outcomes, functional outcomes, and quality of life. In addition, certain measures will be conducted to ensure quality and safety, including centralized photography review and semiannual assessment.

ELIGIBILITY:
Inclusion Criteria:

1. male patients diagnosed with rectal cancer by pathological biopsy;
2. abdominal contrast-enhanced and chest computed tomography (CT) or positron emission tomography-computed tomography (PET-CT) revealed no distal metastasis;
3. Preoperative rectal magnetic resistance (MR) evaluation showed that the tumor was located at or below the peritoneal reflux plane, and at least 1cm above the anal sphincter groove, and did not invade the external anal sphincter;
4. Tumors located above the hiatus of levator ani muscle were evaluated by magnetic resonance imaging as cT1-3, cN0-1, M0, and MRF (-); The tumors located below the hiatus of levator ani muscle were evaluated by magnetic resonance imaging as cT1-2, cN0-1, M0, and MRF (-). After neoadjuvant treatment, the tumor above the hiatus of levator ani muscle is ycT3NxM0 or below; The tumor below the hiatus of levator ani muscle is ycT2NxM0;
5. The patient underwent laparoscopic assisted TME surgery or robotic assisted TME surgery.

Exclusion Criteria:

1. multiple primary cancers;
2. history of open surgery;
3. no preoperative MR evaluation and inadequate evaluation of tumor stage;
4. Patients with rectal cancer who undergo endoscopic resection first and need subsequent transabdominal resection;
5. Pregnant or patients with concomitant inflammatory bowel disease;
6. Patients with preoperative complete bowel obstruction or requiring emergency surgery;
7. Preoperative evaluation indicates that patient may require combined organ resection;
8. Recently receiving treatment for other malignant tumors;
9. Bordeaux type IV low rectal cancer;
10. The preoperative pathological types are signet ring cell carcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, or poorly differentiated carcinoma.

Exit Criteria

1. Refuse surgical treatment after randomization;
2. Open surgery was performed for treatment after randomization;
3. Patients request to withdraw from the study at any time during the entire study process after randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1026 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
intersphincteric resection (ISR) | during the operation
  The primary outcome is the incidence of ISR. ISR is defined according to the definition by a Japanese study group. When the distal resection margin is from dentate line to the intersphincteric groove, ISR will be recorded.The distal resection line of the internal anal sphincter was at the intersphincteric groove in total ISR, between the dentate line and the intersphincteric groove in subtotal ISR and at the dentate line in partial ISR

SECONDARY OUTCOMES:
coloanal anastomosis (CAA) | during the operation
  CAA was defined as the anastomosis of distal colon and surgical anal canal. In CAA anastomosis, the distal resection margin is below the upper level of the levator ani muscle. Conversion to open was defined as an abdominal incision larger than necessary for specimen retrieval.
conversion to open | during the operation
  Conversion to open surgery was defined as an abdominal incision larger than necessary for specimen retrieval extraction.
conversion to transanal TME (TaTME) | during the operation
  Conversion to TaTME was defined as TME that cannot be finished via transabdominal approach, and have to be finished by transanal approach with the help of imaging system and endoscopic instruments. It should be noted that if TME was completely done via transabdominal approach, simply dissecting the internal sphincter and intersphincteric space or finish the coloanal anastomosis via transanal approach were not classified as TaTME
30-day postoperative morbidity | within 30 days after operation
  The 30-day morbidity is defined as intraoperative adverse events and postoperative complications within 30 days. The intraoperative adverse events include intraoperative bleeding (>200 ml), pelvic vascular and nerve injury, vascular injury in other parts, digestive tract injury, ureteral injury, and anastomotic defect. Furthermore, the 30-day postoperative complications are evaluated according to Clavien-Dindo classification
30-day postoperative mortality | within 30 days after operation
  The 30-day mortality is defined as death within 30 day after operation
3-year disease-free survival (DFS) | 3 years after operation
  DFS is defined as the time from randomization to the discovery of local recurrence, distant metastasis, or death of the tumor
3-year local recurrence rate (LR) | 3 years after operation
  LR is defined as tumor recurrence (evaluated by positron emission tomography, computed tomography, or magnetic resistance) that occurs in the pelvic cavity, perineal area, root of inferior mesenteric artery, descending colon, and sigmoid mesenteric area, and is confirmed through pathological biopsy or reoperation.
3-year overall survival (OS) | 3 years after operation
  OS is defined as the time from randomization to death due to any cause.
distance to distal resection margin (DRM) | within 30 days after operation
  The distance to the DRM is defined as the shortest length between the tumor and the DRM. DRM positivity is defined as a distal margin within 1 mm of the tumor.
distance to circumferential resection margin (CRM) | within 30 days after operation
  The distance to the CRM is defined as the shortest length between the tumor and the CRM. CRM positivity is defined as tumor cells within 1 mm from the CRM by microscopy
3-year urinary function | 3 years after operation
  Urinary function will be evaluated by International consultation on incontinence questionnaire short form (ICIQ-SF). The patients will be asked to complete ICIQ-SF every 3 months in the first year after operation, and every 6 months after the first year follow-up, until we finished the 3-year follow-up.
The proportion of patients receiving abdominoperineal resection | during the operation
  the proportion of patients receiving abdominoperineal resection
3-year quality of life | 3 years after operation
  Quality of life will be evaluated by EORTC quality of life questionnaire-core 30 (QLQ-C30) form. The patients will be asked to complete QLQ-C30 every 3 months in the first year after operation, and every 6 months after the first year follow-up, until we finished the 3-year follow-up.
3-year sexual function | 3 years after operation
  Sexual function of male will be evaluated by International Index of Erectile Function (IIEF-5). Sexual function of female will be evaluated by Female Sexual Function Index (FSFI). Evaluation will be performed every 3 months in the first year after operation, and every 6 months after the first year follow-up, until we finished the 3-year follow-up.
3-year defecation function | 3 years after operation
  Defecation function will be evaluated by low anterior resection syndrome (LARS) form. The patients will be asked to complete LARS form every 3 months in the first year after operation, and every 6 months after the first year follow-up, until we finished the 3-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Ph.D., Study Chair — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo Y, He L, Tong W, Chi Z, Ren S, Cui B, Wang Q. A study of intersphincteric resection rate following robotic-assisted total mesorectal excision versus laparoscopic-assisted total mesorectal excision for patients with middle and low rectal cancer: study protocol for a multicenter randomized clinical trial. Trials. 2024 Oct 21;25(1):703. doi: 10.1186/s13063-024-08561-4. PMID 39434171